CLINICAL TRIAL: NCT04969523
Title: Effect of Es-ketamine on Postoperative Delirium Among Old Patients With Lobectomy: a Multicentre, Double-blind, Randomised Clinical Trial
Brief Title: Effect of Es-ketamine on Postoperative Delirium Among Old Patients With Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S001
Record Dates: First submitted 2021-05-19; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- es-ketamine (Experimental): es-ketamine 0.5mg/kg iv
  Interventions: Procedure: lobectomy
- saline (Placebo Comparator): iv saline with the same volume of es-ketamine
  Interventions: Procedure: lobectomy

INTERVENTIONS:
Procedure: lobectomy — Intravenous es-ketamine 0.5mg/kg or saline during lobectomy

SUMMARY:
The purpose of this study is the efficiency of es-ketamine on postoperative delirium among old patients with elective lobectomy

DETAILED DESCRIPTION:
This study aimed to investigate the effect of IV es-ketamine vs saline on the incidence of postoperative delirium. It was hypothesized that IV es-ketamine would reduce the incidence of in-hospital delirium during cardiac surgery lobectomy

ELIGIBILITY:
Inclusion Criteria:

* 60 years old; There is no limit on the gender, ASA (American Society of Anesthesiologists )Ⅰ-Ⅲ

Exclusion Criteria:

* Emergency surgery, severe hepatic and renal dysfunction, shock or coma, psychiatric disease or central nervous system disorder or a history of long-term use of psychiatric medications, cognitive dysfunction, severe arrhythmia or bradycardia, ketamine allergy,drug abuse history and used other sedatives for nearly a week

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Delirium | 7 days after operation
  Confusion Assessment Method (CAM) or CAM-ICU for patients
Postoperative Cognitive Assessment | 7 days after operation
  Montreal Cognitive Assessment

IPD SHARING:
Plan to Share IPD: No